CLINICAL TRIAL: NCT05054283
Title: Baseline Blood Indices as a Marker for Prolonged Length of Hospital Stay in Diabetic Older Patients With Mild or Moderate Covid-19 Infection
Brief Title: Baseline Blood Indices and Prolonged Length of Hospital Stay
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Bilal Katipoglu, Geriatrics, Gulhane Training and Research Hospital
Other Study IDs: 2020-374
Record Dates: First submitted 2021-09-14; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Hospitalism; COVID-19 Pneumonia; Diabetes Mellitus, Type 2
Keywords: Length of hospital stay; Covid-19 Pneumonia; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Length of hospital Stay (normal): The primary outcome was hospital length of stay (LOS), which was calculated according to the number of days of hospitalization. Patients were divided into two groups according to median value of LOS: ≤ 7 days as normal and > 7 days as prolonged LOS.
  Interventions: Diagnostic Test: Inflamatory biomarkers
- Length of hospital Stay (prolonged): The primary outcome was hospital length of stay (LOS), which was calculated according to the number of days of hospitalization. Patients were divided into two groups according to median value of LOS: ≤ 7 days as normal and > 7 days as prolonged LOS.
  Interventions: Diagnostic Test: Inflamatory biomarkers

INTERVENTIONS:
Diagnostic Test: Inflamatory biomarkers — laboratuary parameters of within 24 hours of admission (levels of white blood cell (WBC), lymphocyte neutrophil, hemoglobin (Hb), platelet, fasting glucose, glycated hemoglobin, aspartate aminotransferase (AST) , c-reactive protein (CRP), ferritin, and procalcitonin) were recorded from medical records and collected by two trained fellow geriatricians.

SUMMARY:
During a pandemic, length of hospital stay (LOS) is critical to managing high patient volumes and preserves access to care related to non-COVID-19 for maintaining the healthcare system. Moreover, identiﬁcation of prolonged hospital stay may allow physicians to reevaluate critical patients, focused delivery of specific interventions, and improve the efficiency of hospital care.

Furthermore, in previous recent studies, attention has been paid to patients with diabetes and COVID-19 infection may require a prolonged LOS. However, there is little evidence on prognostic factors associated with an extension of hospitalization in mild or moderate illness due to COVID-19 infection. Therefore, it is crucial to determine the most vulnerable patients with diabetes mellitus even if they have a non-severe COVID-19 infection during the pandemic.

We hypothesize that the clinically relevant inflammatory parameters may have an impact on LOS in older adults with diabetes and non-severe COVID-19 infection. Therefore, we aim to investigate whether baseline inflammatory parameters on admission hospitals as possible predictors of prolonged LOS in older adults with diabetes and non-severe COVID-19 infection during the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* We included all hospitalized Covid-19 patients with diabetes mellitus according to the any established diagnosis prior to admission or American Diabetes Association guidelines for diagnostic criteria

Exclusion Criteria:

* The patients with severe Covid-19 infection, secondary diabetes or type 1 diabetes mellitus were excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The date of hospital admission and discharge of patients and baseline clinical characteristics including age, sex, comorbidities (hypertension, cardiovascular disease, chronic obstructive pulmonary disease and others), diabetes medications (oral anti-diabetic drugs or insulin), and laboratuary parameters of within 24 hours of admission (levels of white blood cell (WBC), lymphocyte neutrophil, hemoglobin (Hb), platelet, fasting glucose, glycated hemoglobin, aspartate aminotransferase (AST) , c-reactive protein (CRP), ferritin, and procalcitonin) were recorded from medical records and collected by two trained fellow geriatricians.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Prolonged Length of hospital | at least 2 week
  The primary outcome was hospital length of stay (LOS), which was calculated according to the number of days of hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane training and research hospital, Ankara, Turkey (Türkiye)